CLINICAL TRIAL: NCT00185016
Title: Women Abuse and the Role of the Family Doctor. Testing an Intervention in a Randomised Controlled Trial.
Brief Title: Women Abuse and the Role of the Family Doctor.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Theia Foundation, Zilveren Kruis Achmea (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: 1,SLFW; Theia 200173
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Improved Recognition of Partner Abuse; Gender Differences in Discussing Partner Abuse; Abused Women's Expectations,Experiences; Abused Women's Health Care Utilisation
Keywords: intimate partner abuse; gender; education; attitude; family doctor; health care utilisation; abused women
MeSH Terms: conditions — Coitus; Behavior

INTERVENTIONS:
Behavioral: a training to improve recognition of partner abuse.

SUMMARY:
The study tested a training to improve recognition of abused female patients in family practice.Effect measures of the training were: number of reported cases wherein the doctor suspected and discussed partner abuse and the number of non-obviuos reasons to suspect partner abuse.We assumed that following a training would improve the recognition of abused women.

Secondary to this trial we explored gender differences of family doctors in discussing partner abuse and we interviewed women recently identified by their family doctor. Medical histories of recently identified abused women were studied to assess health problems and health-care utilisation.

ELIGIBILITY:
Inclusion Criteria:women consulting in family practice, age 18 years and older -

Exclusion Criteria:we excluded only for the interviews: women who were assessed by their family doctor to be in danger because of the abusive situation, women with a psychiatric condition.

-

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Start 2003-03; Study Completion 2004-11

PRIMARY OUTCOMES:
number of reported cases wherein a doctor suspected and discussed partner abuse.

SECONDARY OUTCOMES:
number of cases with non-obvious symptoms wherein a doctor suspected partner abuse.

CONTACTS AND LOCATIONS:
Overall Officials: Toine LM Lagro-Janssen, PhD/MD/FP, Study Chair — Radboud University Medical Centre Nijmegen; Sylvie H Lo Fo Wong, MD/FP, Principal Investigator — Radboud University Medical Centre, Nijmegen
Locations (1):
- Radboud University Medical Centre, Nijmegen, Netherlands